CLINICAL TRIAL: NCT01677546
Title: The Impact of Insulin Pump Bolus Calculator and Wireless Communication With Blood Glucose Meter on Metabolic Control in Children With Type 1 Diabetes Mellitus - Randomised Control Trial
Brief Title: Bolus Calculator and Wireless Communication With Blood Glucose Meter in Management of Type 1 Diabetes Mellitus (T1DM).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Bolus-calculator
Record Dates: First submitted 2012-08-22; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; insulin pump; bolus calculator; Contour Link
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CSII+BC+CL (Experimental): Patients using insulin pump (CSII) bolus calculator (BC) wirelessly connected with blood glucose meter Contour Link (CL)
  Interventions: Device: CSII+BC+CL
- CSII+BC (Experimental): Patients using insulin pump (CSII) bolus calculator (BC) without wireless connection with blood glucose meter (CL)
  Interventions: Device: CSII+BC
- CSII (insulin pump only) (No Intervention): Patients using insulin pump (CSII) without BC and connection with CL

INTERVENTIONS:
Device: CSII+BC+CL — Insulin pump bolus calculator wirelessly communicated with blood glucose meter (Contour Link)
  Other Names: Insulin pump, bolus calculator, bolus Wizard, Contour Link
  Arms: CSII+BC+CL
Device: CSII+BC — Insulin pump bolus calculator without wireless communication with blood glucose meter (Contour Link)
  Other Names: Insulin pump, bolus calculator, bolus Wizard
  Arms: CSII+BC

SUMMARY:
Bolus calculator (BC) is one of the advanced functions in modern insulin pumps (CSII)models. Together with wireless communication with blood glucose meter potentially facilitates achieving the target post prandial glucose levels. In this RCT authors assessed whether use of wireless communication between compatible devices: MiniMed insulin pump and blood glucose meter Contour Link (CL), Bayer results in more frequently bolus calculator using and what is the impact of exerting this tool on metabolic control in type 1 diabetic patients.

DETAILED DESCRIPTION:
In this RCT 156 patients were randomly assigned to one of the 3 arms: group A- subjects using insulin pump bolus calculator wirelessly connected with blood glucose meter, group B- subjects using insulin pump bolus calculator without wireless communication with blood glucose meter or group C- insulin pump, without bolus calculator function. We compared the glycated hemoglobin levels and post- prandial hypoglycaemia after 3 months of observation between the groups. We also assessed secondary endpoints (mentioned above).

Patients were estimated at three time points: at the beginning, after 6 weeks and after 3 months of intervention. Investigators performed computer reports at each visit, with Medtronic CareLink Pro software.

ELIGIBILITY:
Inclusion Criteria:

* 7- 18 years old
* type 1 diabetes mellitus for over 1 year
* treatment with insulin pump with bolus calculator function
* HbA1c < 10%
* expressed written informed consent

Exclusion Criteria:

* recall the consent

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
HbA1c (Glycated hemoglobin) | 3 months

SECONDARY OUTCOMES:
Post- prandial glycaemia | 2 hours after the meals
  Post- prandial glycaemia is express as a mean post- prandial glycaemia counted after the meal consumed between 1- 6 pm during subsequently 7- 10 days
Treatment satisfaction | 3 months
  Simple questions regarded treatment satisfaction and wish to continuation.
Hypoglycaemia episodes and severe hypoglycaemia events | 3 months
  Hypoglycaemia defined as glycaemia below 70 mg/dl and, separately, glycaemia below 50 mg/dl.
Frequency of self- blood glucose monitoring | 3 months
  Number of self- blood glucose monitoring per day
Hyperglycaemic episodes | 3 months
  Hyperglycaemia defined as glycaemia above 180 mg/dl
Frequency of meal boluses | 3 months
  Number of meal boluses per day
Frequency of bolus calculator using | 3 months
  Number of bolus calculator use per day

OTHER OUTCOMES:
Total daily dose of insulin | 3 months
  Total daily dose of insulin express as jm/kg/d
Body mass index- standard deviation (BMI- sds) | 3 months
  Body mass index- sds

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szypowska, A. Professor, Study Chair — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Ramotowska A, Szypowska A. Bolus calculator and wirelessly communicated blood glucose measurement effectively reduce hypoglycaemia in type 1 diabetic children - randomized controlled trial. Diabetes Metab Res Rev. 2014 Feb;30(2):146-53. doi: 10.1002/dmrr.2477. PMID 24115314